CLINICAL TRIAL: NCT01808092
Title: A Phase III, Randomized, Multicentre, Double-blind, Double-dummy, Parallel-group Comparative Study to Determine the Efficacy, Safety And Tolerability of Ceftazidime-Avibactam Versus Meropenem in the Treatment of Nosocomial Pneumonia Including Ventilator-Associated Pneumonia in Hospitalized Adults
Brief Title: A Study Comparing Ceftazidime-Avibactam Versus Meropenem in Hospitalized Adults With Nosocomial Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4281C00001
Record Dates: First submitted 2013-02-28; First posted 2013-03-11 (Estimated); Results first posted 2017-02-03 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Nosocomial Pneumonia (NP); Ventilator-associated Pneumonia (VAP)
Keywords: Ceftazidime,; Meropenem,; Anti-Bacterial Agents,; Anti-Infective Agents,; Therapeutic Uses,; Pharmacologic Actions,; Physiological Effects of Drugs
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated | interventions — Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAZ-AVI (Experimental): Intra-Venous treatment
  Interventions: Drug: ceftazidim-avibactam (CAZ-AVI, experimental product)
- Meropenem (Active Comparator): Intra-Venous treatment
  Interventions: Drug: meropenem (active comparator)

INTERVENTIONS:
Drug: ceftazidim-avibactam (CAZ-AVI, experimental product) — 2000mg ceftazidime plus 500mg avibactam
  Arms: CAZ-AVI
Drug: meropenem (active comparator) — 1000mg of Meropenem
  Arms: Meropenem

SUMMARY:
The purpose of the study is to evaluate the effects of Ceftazidime-Avibactam compared to Meropenem for treating hospitalized adults with nosocomial pneumonia including ventilator-associated pneumonia

DETAILED DESCRIPTION:
A Phase III, Randomized, Multicentre, Double-blind, Double-dummy, Parallel-group Comparative Study to Determine the Efficacy, Safety And Tolerability of Ceftazidime-Avibactam Versus Meropenem in the Treatment of Nosocomial Pneumonia Including Ventilator-Associated Pneumonia in Hospitalized Adults

ELIGIBILITY:
Inclusion Criteria:

* 18 to 90 years of age inclusive
* Females can participate if surgically sterile or completed menopause; if able to have children, must have negative serum pregnancy test, agree not to attempt pregnancy and use acceptable contraception while receiving study therapy and for 1 week after
* Onset of symptoms ≥ 48 hours after admission or <7 days after discharge from an inpatient acute or chronic care facility
* New or worsening infiltrate on chest X-ray obtained within 48 hours prior to randomization
* At least 1 of the following systemic signs:Fever (temperature >38 C) or hypothermia (rectal/core temperature <35 C); White blood cell count >10,000 cells/mm3, or White blood cell count <4500 cells/mm3, or >15% band forms.

Exclusion Criteria:

* Pulmonary disease that, in the investigator's judgment, would preclude evaluation of therapeutic response (e.g. lung cancer, active tuberculosis, cystic fibrosis, granulomatous disease, fungal pulmonary infection or recent pulmonary embolism).
* Patients with lung abscess, pleural empyema or post obstructive pneumonia.
* Patients with an estimated creatinine clearance <16ml/min by Cockcroft Gault formula or patients expected to require haemodialysis or other renal support while on study therapy.
* Acute hepatitis in the prior 6 months, cirrhosis, acute hepatic failure or acute decompensation of chronic hepatic failure.
* Patients receiving hemodialysis or peritoneal dialysis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 969 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chow, MD, FIDSA, Study Director — AstraZeneca
Locations (123):
- Argentina (5):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
  - Research Site, Florida
  - Research Site, La Plata
  - Research Site, Mendoza
- Brazil (4):
  - Research Site, Belo Horizonte
  - Research Site, Campinas/SP
  - Research Site, Curitiba
  - Research Site, São José do Rio Preto
- Bulgaria (4):
  - Research Site, Burgas
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
- China (20):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Jiangyin
  - Research Site, Nanchang
  - Research Site, Qingdao
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Yangzhou
  - Research Site, Zhanjiang
- Czechia (3):
  - Research Site, Kolín
  - Research Site, Kyjov
  - Research Site, Praha 10, Prague
- France (7):
  - Research Site, Limoges
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Strasbourg
  - Research Site, Tours
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Miskolc
  - Research Site, Székesfehérvár
  - Research Site, Veszprém
- India (5):
  - Research Site, Bangalore
  - Research Site, Jaipur
  - Research Site, Lucknow
  - Research Site, Pune
  - Research Site, Varanasi
- Research Site, Bologna, Italy
- Japan (19):
  - Research Site, Fukuoka
  - Research Site, Higashiibaraki-gun
  - Research Site, Ikeda-shi
  - Research Site, Itabashi-ku
  - Research Site, Izumo-shi
  - Research Site, Kagoshima
  - Research Site, Kawasaki-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Kushiro
  - Research Site, Matsuyama
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Sapporo
  - Research Site, Sasebo-shi
  - Research Site, Tsuchiura-shi
  - Research Site, Tsukubo-gun
  - Research Site, Uji-shi
  - Research Site, Uki-shi
  - Research Site, Yanai-shi
- Research Site, Liepāja, Latvia
- Mexico (2):
  - Research Site, Guadalajara
  - Research Site, Monterrey
- Peru (2):
  - Research Site, Cusco
  - Research Site, Lima
- Philippines (2):
  - Research Site, Iloilo City
  - Research Site, Quezon City
- Poland (7):
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Proszowice
  - Research Site, Suwałki
  - Research Site, Łęczna
- Romania (2):
  - Research Site, Craiova
  - Research Site, Timișoara
- Russia (6):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
  - Research Site, Zelenograd
- Research Site, Golnik, Slovenia
- Research Site, Randburg, South Africa
- South Korea (6):
  - Research Site, Ansan-si
  - Research Site, Anyang-si
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Wŏnju
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Sabadell(Barcelona)
  - Research Site, Terrassa (Barcelona)
- Research Site, Taichung, Taiwan
- Research Site, Ankara, Turkey (Türkiye)
- Ukraine (8):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Mykolayiv
  - Research Site, Poltava
  - Research Site, Vinnytsia
- United Kingdom (4):
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Guildford
  - Research Site, Hull
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh

REFERENCES:
- [Derived] Torres A, Wible M, Tawadrous M, Irani P, Stone GG, Quintana A, Debabov D, Burroughs M, Bradford PA, Kollef M. Efficacy and safety of ceftazidime/avibactam in patients with infections caused by beta-lactamase-producing Gram-negative pathogens: a pooled analysis from the Phase 3 clinical trial programme. J Antimicrob Chemother. 2023 Nov 6;78(11):2672-2682. doi: 10.1093/jac/dkad280. PMID 37700689
- [Derived] Cheng K, Newell P, Chow JW, Broadhurst H, Wilson D, Yates K, Wardman A. Safety Profile of Ceftazidime-Avibactam: Pooled Data from the Adult Phase II and Phase III Clinical Trial Programme. Drug Saf. 2020 Aug;43(8):751-766. doi: 10.1007/s40264-020-00934-3. PMID 32602065
- [Derived] Tichy E, Torres A, Bassetti M, Kongnakorn T, Di Virgilio R, Irani P, Charbonneau C. Cost-effectiveness Comparison of Ceftazidime/Avibactam Versus Meropenem in the Empirical Treatment of Hospital-acquired Pneumonia, Including Ventilator-associated Pneumonia, in Italy. Clin Ther. 2020 May;42(5):802-817. doi: 10.1016/j.clinthera.2020.03.014. Epub 2020 Apr 27. PMID 32349879
- [Derived] Stone GG, Bradford PA, Tawadrous M, Taylor D, Cadatal MJ, Chen Z, Chow JW. In Vitro Activity of Ceftazidime-Avibactam against Isolates from Respiratory and Blood Specimens from Patients with Nosocomial Pneumonia, Including Ventilator-Associated Pneumonia, in a Phase 3 Clinical Trial. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02356-19. doi: 10.1128/AAC.02356-19. Print 2020 Apr 21. PMID 32071051
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827
- [Derived] Nichols WW, Stone GG, Newell P, Broadhurst H, Wardman A, MacPherson M, Yates K, Riccobene T, Critchley IA, Das S. Ceftazidime-Avibactam Susceptibility Breakpoints against Enterobacteriaceae and Pseudomonas aeruginosa. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e02590-17. doi: 10.1128/AAC.02590-17. Print 2018 Nov. PMID 30061279
- [Derived] Stone GG, Newell P, Gasink LB, Broadhurst H, Wardman A, Yates K, Chen Z, Song J, Chow JW. Clinical activity of ceftazidime/avibactam against MDR Enterobacteriaceae and Pseudomonas aeruginosa: pooled data from the ceftazidime/avibactam Phase III clinical trial programme. J Antimicrob Chemother. 2018 Sep 1;73(9):2519-2523. doi: 10.1093/jac/dky204. PMID 29912399
- [Derived] Torres A, Zhong N, Pachl J, Timsit JF, Kollef M, Chen Z, Song J, Taylor D, Laud PJ, Stone GG, Chow JW. Ceftazidime-avibactam versus meropenem in nosocomial pneumonia, including ventilator-associated pneumonia (REPROVE): a randomised, double-blind, phase 3 non-inferiority trial. Lancet Infect Dis. 2018 Mar;18(3):285-295. doi: 10.1016/S1473-3099(17)30747-8. Epub 2017 Dec 16. PMID 29254862

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 879 patients were randomized in this study, from 4 geographic regions. The first patient was enrolled on 13 April 2013 and the last patient last visit was on 07 January 2016. Summary tables exclude 62 patients with moderate/severe renal impairment recruited prior to a protocol amendment to the dose regimen for such patients (MSRIBorig).
Pre-assignment Details: The first patient was enrolled on 13 April 2013 and the last patient last vist was on 07 January 2016. Overall, 969 patients were enrolled in this study, 90 of them screen failures.
Groups:
- CAZ-AVI: 2000mg ceftazidime / 500mg avibactam intravenous (IV) infused over 2 hours plus appropriate placebo to meropenem
- Meropenem: meropenem 1000mg IV infused over 30 minutes plus CAZ-AVI placebo
Period: Overall Study
Arm/Group | CAZ-AVI | Meropenem
Started | 409 | 408
Completed | 355 | 363
Not Completed | 54 | 45
Not completed — Death | 39 | 29
Not completed — Lost to Follow-up | 3 | 7
Not completed — Withdrawal by Subject | 9 | 4
Not completed — Other Eligibility criteria | 3 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics analysis is based on safety analysis set: randomized patients who received any amount of study therapy. 9 patients were randomized but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | CAZ-AVI | Meropenem | Total
Number analyzed (Participants) | 405 | 403 | 808
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (16.76) [18 to 89] | 61.7 (17.57) [18 to 90] | 61.7 (17.16) [18 to 90]
Age, Customized [Number; unit: Participants]
  18-45 | 74 | 74 | 148
  46-64 | 124 | 122 | 246
  65-74 | 97 | 95 | 192
  75-90 | 110 | 112 | 222
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 105 | 206
  Male | 304 | 298 | 602
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 226 | 217 | 443
  Black/African American | 3 | 2 | 5
  Native Hawaiian/Pacific Islander | 0 | 0 | 0
  Other | 5 | 7 | 12
  White | 171 | 177 | 348

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Clinical Cure at Test-of-cure (TOC) Visit in the Clinically Modified Intent-to-treat Analysis Set (Co-primary Analyses)
Description: The number of patients meeting the cure criteria: the patient was not a clinical failure at end of treatment and the patient is alive and all signs and symptoms of pneumonia have resolved or improved to an extent that no antibacterial therapy for Nosocomial Pneumonia was taken between end of treatment and test-of-cure inclusive.
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The clinical modified intent-to-treat (cMITT) included all patients who met the minimum disease criteria and received any amount of study treatment, and had either no baseline pathogens or at least one study-qualifying Gram-negative baseline pathogen.
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 356 | 370
participants
  Clinical cure | 245 | 270
  Clinical failure | 79 | 70
  Indeterminate | 32 | 30
Statistical Analysis 1: Comparison: CAZ-AVI vs Meropenem; Statistical analysis for the proportion of patients with clinical cure at TOC in cMITT analysis set; Test type: Non-Inferiority or Equivalence — The statistical test of NI for the primary efficacy analysis will be performed at the 2.5% 1 sided significance level. This test will be based on the lower limit of a 2-sided 95% confidence interval (CI). Consistent with the protocol, NI will be concluded if the lower limit of the 95% CI is greater than -12.5%; p = 0.007, % Risk Difference (RD) — P-value for 1-sided test at test of cure (TOC) with a -12.5% non-inferiority margin, i.e. H0: diff <= -12.5%; RD is CAZ-AVI clinical cure rate minus Meropenem clinical cure rate. The CI was calculated by Miettinen and Nurminen method without adjustment; percentage: units for RD are % = -4.2, 95% CI 2-sided [-10.76 to 2.46]

2. Primary Outcome: The Number of Patients With Clinical Cure at Test-of-cure (TOC) Visit in the Clinically Evaluable at TOC Analysis Set (Co-primary Analyses)
Description: as for outcome 1
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The clinically evaluable (CE) analysis set included all patients in the clinical modified intent-to-treat (cMITT) analysis set who met the stringent criteria for clinical evaluation described in the protocol regarding dosing, prior and concomitant medication, evaluation, etc.
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 257 | 270
participants
  Clinical cure | 199 | 211
  Clinical failure | 58 | 59
Statistical Analysis 1: Comparison: CAZ-AVI vs Meropenem; Statistical analysis for the proportion of patients with clinical cure at TOC in CE at TOC analysis set; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, % Risk Difference (RD) — P-value for 1-sided test at test of cure (TOC) with a -12.5% non-inferiority margin, i.e. H0: diff <= -12.5%; [statistical method as in outcome 1, analysis 1]; percentage: units for RD are % = -0.7, 95% CI 2-sided [-7.86 to 6.39]

3. Secondary Outcome: The Number of Patients With Clinical Cure at Test-of-cure (TOC) Visit in the Microbiologically Modified Intent-to-treat Analysis Set
Description: as for outcome 1
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The microbiological modified intent-to-treat (mMITT) analysis set included all patients who met the minimum disease criteria and received any amount of study treatment, and had at least one study-qualifying Gram-negative baseline pathogen.
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  Clinical cure | 120 | 138
  Clinical failure | 37 | 34
  Indeterminate | 14 | 12

4. Secondary Outcome: The Number of Patients With Clinical Cure at Test-of-cure (TOC) Visit in the Extended Microbiologically Evaluable Analysis Set
Description: as for outcome 1
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The extended-ME (EME) analysis set defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents.
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 125 | 131
participants
  Clinical cure | 96 | 103
  Clinical failure | 29 | 28

5. Secondary Outcome: The Number of Patients With Clinical Cure at Test-of-cure (TOC) Visit in the Microbiologically Evaluable Analysis Set
Description: as for outcome 1
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The microbiologically evaluable (ME) analysis sets defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture that is susceptible to both study agents (CAZ-AVI and meropenem).
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 107 | 118
participants
  Clinical cure | 85 | 94
  Clinical failure | 22 | 24

6. Secondary Outcome: The Number of Patients With Clinical Cure at End of Treatment (EOT) Visit in Microbiologically Modified Intent-to-treat Analysis Set
Description: The number of patients meeting the cure criteria: the patient is alive and all signs and symptoms of pneumonia have resolved or improved such that all antibacterial therapies for Nosocomial Pneumonia are stopped. No antibacterial therapy other than those outlined by the protocol has been administered for Nosocomial Pneumonia prior to end of treatment.
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  Clinical cure | 143 | 161
  Clinical failure | 23 | 18
  Indeterminate | 5 | 5

7. Secondary Outcome: The Number of Patients With Clinical Cure at End of Treatment (EOT) Visit in Clinically Modified Intent-to-treat Analysis Set
Description: as for outcome 6
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 356 | 370
participants
  Clinical cure | 292 | 309
  Clinical failure | 50 | 45
  Indeterminate | 14 | 16

8. Secondary Outcome: The Number of Patients With Clinical Cure at End of Treatment (EOT) Visit in Clinically Evaluable Analysis Set
Description: as for outcome 6
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 291 | 306
participants
  Clinical cure | 253 | 268
  Clinical failure | 38 | 38

9. Secondary Outcome: The Number of Patients With Clinical Cure at End of Treatment (EOT) Visit in Extended Microbiologically Evaluable Analysis Set
Description: as for outcome 6
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 143 | 151
participants
  Clinical cure | 125 | 135
  Clinical failure | 18 | 16

10. Secondary Outcome: The Number of Patients With Clinical Cure at End of Treatment (EOT) Visit in Microbiologically Evaluable Analysis Set
Description: as for outcome 6
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 122 | 138
participants
  Clinical cure | 110 | 126
  Clinical failure | 12 | 12

11. Secondary Outcome: The Number of Patients With a Favorable Per-patient Microbiologic Response at End of Treatment (EOT) Visit in Microbiologically Modified Intent-to-treat Analysis Set
Description: Per-patient "favorable" response indicates that all of the patient's baseline pathogens are "eradicated" or "presumed eradicated". Eradication is defined as: source specimen demonstrates absence of the original baseline pathogen. Presumed eradication is defined as: source specimen was not available to culture and the patient was assessed as a clinical cure.
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  Favorable | 128 | 148
  Unfavorable | 38 | 31
  Indeterminate | 5 | 5

12. Secondary Outcome: The Number of Patients With a Favorable Per-patient Microbiologic Response at Test-of-cure (TOC) Visit in Microbiologically Modified Intent-to-treat Analysis Set
Description: as for outcome 11
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  Favorable | 95 | 118
  Unfavorable | 64 | 54
  Indeterminate | 12 | 12

13. Secondary Outcome: The Number of Patients With a Favorable Per-patient Microbiologic Response at End of Treatment (EOT) Visit in Extended Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 11
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 143 | 151
participants
  Favorable | 112 | 123
  Unfavorable | 31 | 28

14. Secondary Outcome: The Number of Patients With a Favorable Per-patient Microbiologic Response at Test-of-cure (TOC) Visit in Extended Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 11
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 125 | 131
participants
  Favorable | 80 | 89
  Unfavorable | 45 | 42

15. Secondary Outcome: The Number of Patients With a Favorable Per-patient Microbiologic Response at End of Treatment (EOT) Visit in Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 11
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 122 | 138
participants
  Favorable | 96 | 112
  Unfavorable | 26 | 26

16. Secondary Outcome: The Number of Patients With a Favorable Per-patient Microbiologic Response at Test-of-cure (TOC) Visit in Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 11
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 107 | 118
participants
  Favorable | 70 | 83
  Unfavorable | 37 | 35

17. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses at End of Treatment (EOT) Visit in Microbiologically Modified Intent-to-treat Analysis Set at End of Treatment Visit
Description: The number of patients with a favorable per-pathogen microbiological response: favorable microbiological response includes: Eradication where, source specimen demonstrates absence of the original baseline pathogen. Presumed eradication where, source specimen was not available to culture and the patient was assessed as a clinical cure.
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The microbiological modified intent-to-treat (mMITT) analysis set included all patients who met the minimum disease criteria and received any amount of study treatment, and had at least one study-qualifying Gram-negative baseline pathogen. (pathogens in ≥10 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants with favorable responses
  Enterobacter aerogenes (n=8, 8) | 6 | 5
  Enterobacter cloacae (n=26, 22) | 25 | 20
  Escherichia coli (n=17, 20) | 15 | 18
  Klebsiella pneumoniae (n=59, 71) | 49 | 65
  Proteus mirabilis (n=14, 12) | 12 | 10
  Serratia marcescens (n=15, 13) | 12 | 11
  Haemophilus influenzae (n=16, 25) | 15 | 25
  Pseudomonas aeruginosa (n=58, 47) | 33 | 27
  Staphylococcus aureus (n=24, 34) | 21 | 32

18. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses at End of Treatment (EOT) Visit in Extended Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 17
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The extended-ME (EME) analysis set defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents. (pathogens in ≥10 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 143 | 151
participants with favorable responses
  Enterobacter aerogenes (n=6, 7) | 4 | 5
  Enterobacter cloacae (n=22, 17) | 22 | 17
  Escherichia coli (n=14, 18) | 13 | 17
  Klebsiella pneumoniae (n=46, 57) | 39 | 53
  Proteus mirabilis (n=9, 8) | 8 | 6
  Serratia marcescens (n=13, 10) | 12 | 8
  Haemophilus influenzae (n=14, 16) | 14 | 16
  Pseudomonas aeruginosa (n=50, 41) | 30 | 24
  Staphylococcus aureus (n=18, 26) | 16 | 25

19. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses at End of Treatment (EOT) Visit in Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 17
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The microbiologically evaluable (ME) analysis sets defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture that is susceptible to both study agents (CAZ-AVI and meropenem). (pathogens in ≥10 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 122 | 138
participants with favorable responses
  Enterobacter aerogenes (n=6, 7) | 4 | 5
  Enterobacter cloacae (n=22, 17) | 22 | 17
  Escherichia coli (n=13, 18) | 13 | 17
  Klebsiella pneumoniae (n=45, 55) | 38 | 51
  Proteus mirabilis (n=9, 8) | 8 | 6
  Serratia marcescens (n=13, 10) | 12 | 8
  Haemophilus influenzae (n=12, 15) | 12 | 15
  Pseudomonas aeruginosa (n=38, 34) | 22 | 19
  Staphylococcus aureus (n=16, 23) | 14 | 22

20. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses at Test-of-cure (TOC) Visit in Microbiologically Modified Intent-to-treat Analysis Set at Test-of-cure Visit
Description: as for outcome 17
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 17
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants with favorable responses
  Enterobacter aerogenes (n=8, 8) | 5 | 5
  Enterobacter cloacae (n=26, 22) | 21 | 13
  Escherichia coli (n=17, 20) | 13 | 16
  Klebsiella pneumoniae (n=59, 71) | 37 | 53
  Proteus mirabilis (n=14, 12) | 11 | 8
  Serratia marcescens (n=15, 13) | 10 | 8
  Haemophilus influenzae (n=16, 25) | 14 | 23
  Pseudomonas aeruginosa (n=58, 47) | 22 | 18
  Staphylococcus aureus (n=24, 34) | 11 | 25

21. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses at Test-of-cure (TOC) Visit in Extended Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 17
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 18
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 125 | 131
participants with favorable responses
  Enterobacter aerogenes (n=6, 5) | 5 | 3
  Enterobacter cloacae (n=21, 11) | 18 | 7
  Escherichia coli (n=11, 18) | 10 | 16
  Klebsiella pneumoniae (n=37, 49) | 29 | 39
  Proteus mirabilis (n=11, 8) | 9 | 6
  Serratia marcescens (n=12, 8) | 9 | 5
  Haemophilus influenzae (n=11, 13) | 11 | 12
  Pseudomonas aeruginosa (n=42, 35) | 18 | 14
  Staphylococcus aureus (n=14, 22) | 5 | 17

22. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses at Test-of-cure (TOC) Visit in Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 17
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 19
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 107 | 118
participants with favorable responses
  Enterobacter aerogenes (n=6, 5) | 5 | 3
  Enterobacter cloacae (n=21, 11) | 18 | 7
  Escherichia coli (n=10, 18) | 10 | 16
  Klebsiella pneumoniae (n=37, 47) | 29 | 38
  Proteus mirabilis (n=11, 8) | 9 | 6
  Serratia marcescens (n=12, 8) | 9 | 5
  Haemophilus influenzae (n=9, 12) | 9 | 11
  Pseudomonas aeruginosa (n=31, 28) | 13 | 12
  Staphylococcus aureus (n=13, 19) | 4 | 15

23. Secondary Outcome: The Number of Patients With Clinical Cure in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Clinically Modified Intent-to-treat Analysis Set at End of Treatment Visit
Description: as for outcome 6
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The microbiological modified intent-to-treat (mMITT) analysis set included all patients who met the minimum disease criteria and received any amount of study treatment, and had at least one study-qualifying Gram-negative baseline pathogen. (pathogens in ≥5 patients)
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  All (n=45, 54) | 40 | 45
  Enterobacteriaceae (n=34, 41) | 32 | 33
  Enterobacter aerogenes (n=4, 2) | 3 | 2
  Enterobacter cloacae (n=6, 6) | 6 | 4
  Escherichia coli (n=6, 5) | 5 | 3
  Klebsiella pneumoniae (n=20, 30) | 20 | 26
  Gram- pathogens not Enterobacteriaceae (n=11,16) | 8 | 14
  Pseudomonas aeruginosa (n=11, 15) | 8 | 13

24. Secondary Outcome: The Number of Patients With Clinical Cure in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Clinically Evaluable at End of Treatment Analysis Set
Description: as for outcome 6
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The clinically evaluable (CE) analysis set included all patients in the clinical modified intent-to-treat (cMITT) analysis set who met the stringent criteria for clinical evaluation described in the protocol regarding dosing, prior and concomitant medication, evaluation, etc. (pathogens in ≥5 patients)
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 291 | 306
participants
  All (n=39, 49) | 35 | 42
  Enterobacteriaceae (n=29, 37) | 27 | 31
  Enterobacter aerogenes (n=4, 2) | 3 | 2
  Enterobacter cloacae (n=6, 5) | 6 | 3
  Escherichia coli (n=6, 4) | 5 | 3
  Klebsiella pneumoniae (n=16, 28) | 16 | 25
  Gram- pathogens not Enterobacteriaceae (n=10,14) | 8 | 13
  Pseudomonas aeruginosa (n=10, 13) | 8 | 12

25. Secondary Outcome: The Number of Patients With Clinical Cure in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 6
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The microbiologically evaluable (ME) analysis sets defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture that is susceptible to both study agents (CAZ-AVI and meropenem). (pathogens in ≥5 patients)
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 122 | 138
participants
  All (n=32, 40) | 31 | 36
  Enterobacteriaceae (n=28, 35) | 27 | 31
  Enterobacter aerogenes (n=4, 2) | 3 | 2
  Enterobacter cloacae (n=6, 5) | 6 | 3
  Escherichia coli (n=5, 4) | 5 | 3
  Klebsiella pneumoniae (n=16, 26) | 16 | 25
  Gram- pathogens not Enterobacteriaceae (n=4,7) | 4 | 7
  Pseudomonas aeruginosa (n=4, 6) | 4 | 6

26. Secondary Outcome: The Number of Patients With Clinical Cure in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Clinically Modified Intent-to-treat Analysis Set at Test-of-cure Visit
Description: as for outcome 1
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  All (n=45, 54) | 35 | 40
  Enterobacteriaceae (n=34, 41) | 28 | 29
  Enterobacter aerogenes (n=4, 2) | 3 | 2
  Enterobacter cloacae (n=6, 6) | 6 | 4
  Escherichia coli (n=6, 5) | 4 | 3
  Klebsiella pneumoniae (n=20, 30) | 16 | 22
  Gram- pathogens not Enterobacteriaceae (n=11,16) | 7 | 13
  Pseudomonas aeruginosa (n=11, 15) | 7 | 13

27. Secondary Outcome: The Number of Patients With Clinical Cure in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Clinically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 1
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 257 | 270
participants
  All (n=36, 41) | 29 | 32
  Enterobacteriaceae (n=27, 30) | 23 | 22
  Enterobacter cloacae (n=5, 5) | 5 | 3
  Escherichia coli (n=5, 4) | 4 | 3
  Klebsiella pneumoniae (n=14, 22) | 12 | 17
  Gram- pathogens not Enterobacteriaceae (n=9,13) | 6 | 12
  Pseudomonas aeruginosa (n=9, 13) | 6 | 12

28. Secondary Outcome: The Number of Patients With Clinical Cure in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 1
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 25
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 107 | 118
participants
  All (n=29, 32) | 25 | 26
  Enterobacteriaceae (n=26, 28) | 23 | 22
  Enterobacter cloacae (n=5, 5) | 5 | 3
  Escherichia coli (n=4, 4) | 4 | 3
  Klebsiella pneumoniae (n=14, 20) | 12 | 17
  Gram- pathogens not Enterobacteriaceae (n=3,6) | 2 | 6
  Pseudomonas aeruginosa (n=3, 6) | 2 | 6

29. Secondary Outcome: Number of Patients With a Favorable Per-patient Microbiologic Response in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Microbiologically Modified Intent-to-treat Analysis Set at End of Treatment Visit
Description: as for outcome 11
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The microbiological modified intent-to-treat (mMITT) analysis set included all patients who met the minimum disease criteria and received any amount of study treatment, and had at least one study-qualifying Gram-negative baseline pathogen. Patients infected with ceftazidime-resistant Gram negative pathogens at EOT
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 46 | 54
participants
  Favorable | 35 | 39
  Unfavorable | 10 | 13
  Indeterminate | 1 | 2

30. Secondary Outcome: Number of Patients With a Favorable Per-patient Microbiologic Response in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Extended Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 11
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The extended-ME (EME) analysis set defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents. Patients infected with ceftazidime-resistant Gram negative pathogens at EOT
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 40 | 49
participants
  Favorable | 31 | 36
  Unfavorable | 9 | 13

31. Secondary Outcome: Number of Patients With a Favorable Per-patient Microbiologic Response in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 11
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The microbiologically evaluable (ME) analysis sets defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture that is susceptible to both study agents (CAZ-AVI and meropenem). Patients infected with ceftazidime-resistant Gram negative pathogens at EOT
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 33 | 40
participants
  Favorable | 26 | 29
  Unfavorable | 7 | 11

32. Secondary Outcome: Number of Patients With a Favorable Per-patient Microbiologic Response in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Microbiologically Modified Intent-to-treat Analysis Set at Test-of-cure Visit
Description: as for outcome 11
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The microbiological modified intent-to-treat (mMITT) analysis set included all patients who met the minimum disease criteria and received any amount of study treatment, and had at least one study-qualifying Gram-negative baseline pathogen. Patients infected with ceftazidime-resistant Gram negative pathogens at TOC
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 46 | 54
participants
  Favorable | 27 | 27
  Unfavorable | 16 | 23
  Indeterminate | 3 | 4

33. Secondary Outcome: Number of Patients With a Favorable Per-patient Microbiologic Response in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Extended Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 11
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The extended-ME (EME) analysis set defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents. Patients infected with ceftazidime-resistant Gram negative pathogens at TOC
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 37 | 41
participants
  Favorable | 23 | 21
  Unfavorable | 14 | 20

34. Secondary Outcome: Number of Patients With a Favorable Per-patient Microbiologic Response in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 11
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The microbiologically evaluable (ME) analysis sets defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture that is susceptible to both study agents (CAZ-AVI and meropenem). Patients infected with ceftazidime-resistant Gram negative pathogens at TOC
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 30 | 32
participants
  Favorable | 21 | 18
  Unfavorable | 9 | 14

35. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Microbiologically Modified Intent-to-treat Analysis Set at End of Treatment Visit
Description: as for outcome 17
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The microbiological modified intent-to-treat (mMITT) analysis set included all patients who met the minimum disease criteria and received any amount of study treatment, and had at least one study-qualifying Gram-negative baseline pathogen. Patients infected with ceftazidime-resistant Gram negative pathogens at EOT (pathogens in ≥5 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 46 | 54
participants with favorable responses
  Enterobacter aerogenes (n=4, 2) | 3 | 2
  Enterobacter cloacae (n=6, 6) | 6 | 6
  Escherichia coli (n=6, 5) | 5 | 4
  Klebsiella pneumoniae (n=20, 30) | 18 | 26
  Pseudomonas aeruginosa (n=11, 15) | 8 | 7

36. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Extended Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 17
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: The extended-ME (EME) analysis set defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents. Patients infected with ceftazidime-resistant Gram negative pathogens at EOT (pathogens in ≥5 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 40 | 49
participants with favorable responses
  Enterobacter aerogenes (n=4, 2) | 3 | 2
  Enterobacter cloacae (n=6, 5) | 6 | 5
  Escherichia coli (n=6, 4) | 5 | 4
  Klebsiella pneumoniae (n=16, 28) | 14 | 25
  Pseudomonas aeruginosa (n=10, 13) | 8 | 6

37. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses in Patients With Pathogens Resistant to Ceftazidime at End of Treatment (EOT) Visit in Microbiologically Evaluable at End of Treatment Analysis Set
Description: as for outcome 17
Time Frame: Patients were followed after the last IV dose but no later than 24 hours after the last IV dose.
Population: Microbiologically evaluable (ME) analysis sets defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture that is susceptible to both study agents (CAZ-AVI and meropenem). Patients infected with ceftazidime-resistant Gram negative pathogens at EOT (pathogens in ≥5 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 33 | 40
participants with favorable responses
  Enterobacter aerogenes (n=4, 2) | 3 | 2
  Enterobacter cloacae (n=6, 5) | 6 | 5
  Escherichia coli (n=5, 4) | 5 | 4
  Klebsiella pneumoniae (n=16, 26) | 14 | 23
  Pseudomonas aeruginosa (n=4, 6) | 3 | 1

38. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Microbiologically Modified Intent-to-treat Analysis Set at Test-of-cure Visit
Description: as for outcome 17
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The microbiological modified intent-to-treat (mMITT) analysis set included all patients who met the minimum disease criteria and received any amount of study treatment, and had at least one study-qualifying Gram-negative baseline pathogen. Patients infected with ceftazidime-resistant Gram negative pathogens at TOC (pathogens in ≥5 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 46 | 54
participants with favorable responses
  Enterobacter aerogenes (n=4, 2) | 3 | 2
  Enterobacter cloacae (n=6, 6) | 5 | 5
  Escherichia coli (n=6, 5) | 4 | 4
  Klebsiella pneumoniae (n=20, 30) | 15 | 18
  Pseudomonas aeruginosa (n=11, 15) | 4 | 4

39. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Extended Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 17
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: The extended-ME (EME) analysis set defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture regardless of susceptibility to study agents. Patients infected with ceftazidime-resistant Gram negative pathogens at TOC (pathogens in ≥5 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 37 | 41
participants with favorable responses
  Enterobacter cloacae (n=5, 5) | 4 | 4
  Escherichia coli (n=5, 4) | 4 | 4
  Klebsiella pneumoniae (n=14, 22) | 11 | 14
  Pseudomonas aeruginosa (n=9, 13) | 3 | 3

40. Secondary Outcome: The Number of Favorable Per-pathogen Microbiologic Responses in Patients With Pathogens Resistant to Ceftazidime at Test-of-cure (TOC) Visit in Microbiologically Evaluable at Test-of-cure Analysis Set
Description: as for outcome 17
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: Microbiologically evaluable (ME) analysis sets defined as all patients in clinically evaluable (CE) analysis set with at least 1 etiologic pathogen from an adequate baseline culture that is susceptible to both study agents (CAZ-AVI and meropenem). Patients infected with ceftazidime-resistant Gram negative pathogens at TOC (pathogens in ≥5 patients)
Measure: Number; unit: participants with favorable responses
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 30 | 32
participants with favorable responses
  Enterobacter cloacae (n=5, 5) | 4 | 4
  Escherichia coli (n=4, 4) | 4 | 4
  Klebsiella pneumoniae (n=14, 20) | 11 | 13
  Pseudomonas aeruginosa (n=3, 6) | 1 | 1

41. Secondary Outcome: The Number of Patients With Death Due to Any Cause (All-cause Mortality) at Test-of-cure (TOC) Visit in Microbiologically Modified Intent-to-treat Analysis Set at Test-of-cure Visit
Description: The number of patients with death due to any cause (all-cause mortality) in microbiologically modified intent-to-treat analysis set at test-of-cure visit.
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  Number of patients who died (all cause mortality) | 16 | 14
  Deaths due to disease progression | 6 | 5
  Number of patients with any AE with outcome=death | 10 | 9
  Number of patients alive | 153 | 170
  Number of patients with unknown survival status | 2 | 0

42. Secondary Outcome: The Number of Patients With Death Due to Any Cause (All-cause Mortality) at Test-of-cure (TOC) Visit in Clinically Modified Intent-to-treat Analysis Set at Test-of-cure Visit
Description: The number of patients with death due to any cause (all-cause mortality) in clinically modified intent-to-treat analysis set at test-of-cure visit.
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 356 | 370
participants
  Number of patients who died (all cause mortality) | 29 | 25
  Deaths due to disease progression | 10 | 6
  Number of patients with any AE with outcome=death | 19 | 19
  Number of patients alive | 316 | 341
  Number of patients with unknown survival status | 11 | 4

43. Secondary Outcome: The Number of Patients With Death Due to Any Cause (All-cause Mortality) at Test-of-cure (TOC) Visit in the Clinically Evaluable at Test-of-cure Analysis Set
Description: The number of patients with death due to any cause (all-cause mortality) in the clinically evaluable at test-of-cure analysis set.
Time Frame: At the test-of-cure (TOC) visit (Day 21 to 25)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 257 | 270
participants
  Number of patients who died (all cause mortality) | 11 | 8
  Deaths due to disease progression | 5 | 4
  Number of patients with any AE with outcome=death | 6 | 4
  Number of patients alive | 245 | 262
  Number of patients with unknown survival status | 1 | 0

44. Secondary Outcome: The Number of Patients With Death Due to Any Cause (All-cause Mortality) in Microbiologically Modified Intent-to-treat Analysis Set at Day 28
Description: The number of patients with death due to any cause (all-cause mortality) in microbiologically modified intent-to-treat analysis set at day 28.
Time Frame: at Day 28 from randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  Number of patients who died (all cause mortality) | 17 | 16
  Deaths due to disease progression | 6 | 5
  Number of patients with any AE with outcome=death | 11 | 11
  Number of patients alive | 152 | 168
  Number of patients with unknown survival status | 2 | 0

45. Secondary Outcome: The Number of Patients With Death Due to Any Cause (All-cause Mortality) in Clinically Modified Intent-to-treat Analysis Set at Day 28
Description: The number of patients with death due to any cause (all-cause mortality) in clinically modified intent-to-treat analysis set at day 28.
Time Frame: at Day 28 from randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 356 | 370
participants
  Number of patients who died (all cause mortality) | 30 | 27
  Deaths due to disease progression | 10 | 6
  Number of patients with any AE with outcome=death | 20 | 21
  Number of patients alive | 315 | 339
  Number of patients with unknown survival status | 11 | 4

46. Secondary Outcome: The Number of Patients With Death Due to Any Cause (All-cause Mortality) in the Clinically Evaluable at Test-of-cure Analysis Set at Day 28
Description: The number of patients with death due to any cause (all-cause mortality) in the clinically evaluable at test-of-cure analysis set at day 28.
Time Frame: at Day 28 from randomization
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 257 | 270
participants
  Number of patients who died (all cause mortality) | 12 | 9
  Deaths due to disease progression | 5 | 4
  Number of patients with any AE with outcome=death | 7 | 5
  Number of patients alive | 244 | 261
  Number of patients with unknown survival status | 1 | 0

47. Secondary Outcome: The Number of Patients Discharged From Hospital up to Test-of-cure (TOC) Visit in Microbiologically Modified Intent-to-treat Analysis Set
Description: The number of patients discharged from hospital in microbiologically modified intent-to-treat analysis set.
Time Frame: up to 25 days from randomization
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 171 | 184
participants
  Number of patients with admission date | 170 | 182
  Number of patients with at least one discharge | 71 | 75
  1 discharge | 71 | 74
  2 discharges | 0 | 1
  >2 discharges | 0 | 0

48. Secondary Outcome: The Number of Patients Discharged From Hospital up to Test-of-cure (TOC) Visit in the Clinically Modified Intent-to-treat Analysis Set
Description: The number of patients discharged from hospital in the clinically modified intent-to-treat analysis set.
Time Frame: up to 25 days from randomization
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 356 | 370
participants
  Number of patients with admission date | 355 | 366
  Number of patients with at least one discharge | 206 | 206
  1 discharge | 201 | 200
  2 discharges | 5 | 4
  >2 discharges | 0 | 2

49. Secondary Outcome: The Number of Patients Discharged From Hospital up to Test-of-cure (TOC) Visit in the Clinically Evaluable at Test-of-cure Analysis Set
Description: The number of patients discharged from hospital in the clinically evaluable at test-of-cure analysis set.
Time Frame: up to 25 days from randomization
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | CAZ-AVI | Meropenem
Number analyzed (Participants) | 257 | 270
participants
  Number of patients with admission date | 256 | 266
  Number of patients with at least one discharge | 148 | 155
  1 discharge | 144 | 151
  2 discharges | 4 | 3
  >2 discharges | 0 | 1

ADVERSE EVENTS:
Time Frame: Nonserious AEs and SAEs are collected for each patient from date when informed consent is obtained until the date of final protocol follow-up, study withdrawal or date of death from any cause, whichever came first, assessed up to 28 days.
Description: AEs spontaneously reported by the patient or care provider or reported in response to open question from the study center personnel, or revealed by observation were to be collected and recorded in the eCRF. Summary tables include all randomized patients but 62 MSRIBorig patients and 9 patients who didn't receive study treatment after randomization.
Arm/Group | CAZ-AVI | Meropenem
Serious Adverse Events (participants affected / at risk) | 75/405 | 54/403
Other Adverse Events (participants affected / at risk) | 198/405 | 195/403
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAZ-AVI (N=405) | Meropenem (N=403)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (3) | 3 (4)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (4) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 3 (3) | 1 (1)
Intentional medical device removal by patient (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Subacute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
CNS ventriculitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 2 (2)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 1 (1) | 0 (0)
HIV infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 6 (6)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 4 (5)
Septic shock (Infections and infestations) | 3 (3) | 3 (3)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weaning failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Brachial plexopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchoplegia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CAZ-AVI (N=405) | Meropenem (N=403)
Anaemia (Blood and lymphatic system disorders) | 24 (25) | 18 (21)
Abdominal pain (Gastrointestinal disorders) | 10 (11) | 8 (8)
Constipation (Gastrointestinal disorders) | 25 (25) | 31 (38)
Diarrhoea (Gastrointestinal disorders) | 60 (65) | 62 (68)
Nausea (Gastrointestinal disorders) | 13 (13) | 7 (7)
Vomiting (Gastrointestinal disorders) | 23 (28) | 22 (24)
Oedema peripheral (General disorders) | 17 (18) | 15 (15)
Pyrexia (General disorders) | 10 (11) | 13 (20)
Urinary tract infection (Infections and infestations) | 11 (11) | 14 (14)
Alanine aminotransferase increased (Investigations) | 16 (16) | 19 (20)
Aspartate aminotransferase increased (Investigations) | 16 (16) | 17 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 43 (47) | 33 (40)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (10) | 6 (6)
Insomnia (Psychiatric disorders) | 4 (4) | 11 (11)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 7 (7)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 9 (13) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 13 (13)
Hypertension (Vascular disorders) | 14 (14) | 15 (16)
Hypotension (Vascular disorders) | 10 (10) | 8 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No